CLINICAL TRIAL: NCT03071653
Title: Left Cardiac Sympathetic Denervation (LCSD) for Cardiomyopathy Feasibility Pilot Study
Brief Title: Left Cardiac Sympathetic Denervation for Cardiomyopathy Feasibility Pilot Study
Acronym: LCSD
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: COVID and Funding
Sponsor: University of Cape Town (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Mpiko Ntsekhe, Professor, University of Cape Town
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 001001001
Record Dates: First submitted 2017-02-24; First posted 2017-03-07 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Dilated Cardiomyopathy; Ischemic Cardiomyopathy; Non-ischemic Cardiomyopathy
Keywords: Cardiomyopathy; Left Cardiac Sympathetic Denervation
MeSH Terms: conditions — Cardiomyopathy, Dilated; Cardiomyopathies

STUDY DESIGN:
Intervention Model Description: Randomised Control Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Left Cardiac Sympathetic Denervation (LCSD) (Active Comparator): Left Cardiac Sympathetic Denervation (LCSD) in addition to Optimal Medical Therapy (OMT)
  Interventions: Procedure: Left Cardiac Sympathetic Denervation (LCSD); Other: Optimal Medical Therapy
- OMT only (Other): Optimal Medical Therapy (OMT) only
  Interventions: Other: Optimal Medical Therapy

INTERVENTIONS:
Procedure: Left Cardiac Sympathetic Denervation (LCSD) — The procedure involves the surgical removal of the lower half of the left stellate ganglion (T1) and thoracic ganglia (T2-T4), thereby removing the pro-arrhythmic noradrenergic input to the ventricles
  Arms: Left Cardiac Sympathetic Denervation (LCSD)
Other: Optimal Medical Therapy — All eligible patients with heart failure and depressed left ventricular systolic function will receive guideline and evidence based optimal tolerated medical therapy. The level of risk associated with optimal medical therapy is considered very low. For the majority of patients with heart failure and depressed left ventricular systolic function this will include:
  1. A renin angiotensin system blocker at highest tolerated doses (e.g., enalapril 10mg twice daily or equivalent)
  2. A mineralocorticoid receptor antagonist (e.g., Spironolactone 25-50mg daily or equivalent)
  3. A Beta-blocker (e.g., Carvedilol 25mg twice daily or equivalent)
  4. The use of a loop diuretic and digitalis will be clinically driven and used at the discretion of the attending clinician

SUMMARY:
A randomized controlled trial to test the potential safety and efficacy of LCSD in patients with heart failure due to non-ischemic and ischemic cardiomyopathy at the University of Cape Town. Left Cardiac Sympathetic Denervation (LCSD) is a surgical intervention that modulates the autonomic innervation of the cardiac system. This is important because: a] sympathetic and parasympathetic tone has a profound effect on the threshold for ventricular tachyarrhythmias-the main cause of sudden cardiac death in this population; and b] autonomic dysfunction (which is characterized by an imbalance between sympathetic and parasympathetic activation), plays an important detrimental role in the pathophysiology and progression of heart failure.

DETAILED DESCRIPTION:
STUDY SUMMARY

TITLE Left Cardiac Sympathetic Denervation (LCSD) for Cardiomyopathy Study DESIGN Phase II feasibility parallel randomised controlled trial (RCT) AIMS Assess the feasibility and safety of LCSD in patients with cardiomyopathy and heart failure OUTCOME MEASURES Recruitment rates, retention, follow-up and safety POPULATION 30 patients with heart failure secondary to cardiomyopathy ELIGIBILITY Adult participants with ischemic and non-ischemic cardiomyopathy DURATION 18 months follow up

METHODS:

Participants will be randomized to receive LCSD in addition to optimal medical therapy in the intervention arm (15 patients) and optimal medical therapy in the active control arm (15 patients). Participants would be recruited from both inpatient and outpatient general medical and cardiology wards and clinics at Groote Schuur Hospital where patients with the syndrome of heart failure are frequently referred for subspecialty evaluation and management. Eligible patients who meet the inclusion criteria would be randomized to undergo LCSD in addition to optimal medical therapy (intervention arm) or receive standard optimal medical therapy (active placebo). Optimal therapy for patients with cardiomyopathy and heart failure currently consists of an ace-inhibitor or angiotensinogen receptor blocker, beta-blocker, mineralocorticoid receptor antagonist with or without a loop diuretic, and digoxin. All patients in the study would receive an implantable loop recorder to allow for the accurate determination of episodes of symptomatic and asymptomatic ventricular tachyarrhythmias. In order not to lose all of the clinical outcome information obtained in the pilot phase of the study, we would propose only assessing the pre-specified feasibility and safety aspects of the study and keeping the data on efficacy outcomes blinded for inclusion in the fully powered main study.

The LCSD procedure The procedure involves the surgical removal of the lower half of the left stellate ganglion (T1) and thoracic ganglia (T2-T4), thereby removing the pro-arrhythmic noradrenergic input to the ventricles (3). LCSD raises the ventricular fibrillation threshold without impairing cardiac contractility or reducing heart rate. LCSD results in pre-ganglionic denervation, thus preventing re-innervation and producing permanent antifibrillatory effects. This procedure can be performed by video-assisted thoracoscopic surgery (VATS) usually in less than 45 minutes and will be conducted by thoracic surgeons at Groote Schuur Hospital. The lead thoracic surgeon (J.R.) has a large experience in performing this procedure for the indication of hyperhidrosis in over 200 patients (personal communication). This experienced thoracic surgeon will lead a team of thoracic surgeons (T.P., L.M.) to perform the procedure.

Implantable loop recorder (ILR) insertion The implantable loop recorder is a small device that will be inserted at the end of the LCSD procedure by the thoracic surgeon or after enrolment in the optimal medical therapy arm by a cardiologist. This loop recorder is inserted under sterile conditions in the catheter laboratory or operating theatre. In the catheter laboratory, the device is inserted under local anaesthetic, subcutaneously over the left precordium and usually takes less than 15 minutes. The implantable loop recorder is a well-established device to quantify and detect atrial and ventricular tachyarrhythmias with an excellent safety record. The device has a battery life of up to 3 years and can be removed via a small skin incision at the end of the study. Implantable loop recorder insertion does not carry risk of known major complications. There is a minimal risk (<1%) of complications (infection, bleeding) as the device is implanted subcutaneously. Potential complications include superficial skin infections that readily responds to antibiotics. Device removal is easy to perform and is seldom required.

Optimal Medical Therapy

All eligible patients with heart failure and depressed left ventricular systolic function will receive guideline and evidence based optimal tolerated medical therapy. The level of risk associated with optimal medical therapy is considered very low. For the majority of patients with heart failure and depressed left ventricular systolic function this will include:

1. A renin angiotensin system blocker at highest tolerated doses (e.g., enalapril 10mg twice daily or equivalent)
2. A mineralocorticoid receptor antagonist (e.g., Spironolactone 25-50mg daily or equivalent)
3. A Beta-blocker (e.g., Carvedilol 25mg twice daily or equivalent)
4. The use of a loop diuretic and digitalis will be clinically driven and used at the discretion of the attending clinician

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* New York Heart Association (NYHA) II/III stable heart failure due to an ischemic or non-ischemic cardiomyopathy with a Left Ventricular Ejection Fraction <=35% based on Echocardiogram, ERNA or MRI performed in the last 12 months. For the purpose of this study, Ischemic cardiomyopathy will be defined as Left Ventricular systolic dysfunction (Ejection Fraction <35%) associated with 75% narrowing of at least 1 of the 3 major coronary arteries, a documented history of a ST elevation myocardial infarction or significant regional wall motion abnormality on an echocardiogram. Non-ischemic cardiomyopathy will be defined as Left Ventricular systolic dysfunction <35% in the absence of known coronary artery disease or regional wall motion abnormality on echocardiography.
* No history of a prior cardiac arrest or sustained (>30 seconds or <30s if haemodynamically unstable) ventricular tachyarrhythmia.
* Signed informed consent forms will be available in IsiXhosa, Afrikaans and English.

Exclusion Criteria:

* History of prior unexplained syncope, sudden cardiac arrest or ventricular arrhythmia
* Peripartum cardiomyopathy or cardiomyopathy associated with thyrotoxicosis
* History of coronary revascularization or percutaneous intervention in the preceding 3 months
* Myocardial infarction in the preceding 1 month
* NYHA IV at enrollment
* Patient taking an antiarrhythmic drug (not including beta-blockers)
* Pregnancy
* Any non-cardiac condition that is associated with a high likelihood of death during the trial such as major organ dysfunction or malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-11-24 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recruiting | 36 months
  Recruitment rate
Feasibility of performing the procedure in recruited patients | 36 months
  Patient retention
Procedure related complications | 36 months
  Measured by:• Horner's syndrome in those under going LCSD • Pneumothorax in those undergoing LCSD • Implantable loop recorder site sepsis

SECONDARY OUTCOMES:
Mortality and morbidity | 36 months
  Measured by: All cause mortality; Heart failure related mortality; Hospital admissions; Ventricular arrhythmias;
Functional capacity: Measured by 6 minute walk test Quality of life at 6 months Admission to hospital for heart failure Functional Capacity | 6 monthly for 36 months
  Measured by 6 minute walk test
Functional capacity: Quality of life (EQ-5D questionnaire) Quality of life at 6 months Admission to hospital for heart failure Functional Capacity | 6 monthly for 36 months
  Quality of life (EQ-5D questionnaire)
End Systolic and Diastolic volumes | 6 monthly for 36 months
  End Systolic and Diastolic volumes as determined by Echocardiography

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cape Town, Cape Town, Western Cape, South Africa